CLINICAL TRIAL: NCT04363762
Title: An Internet-based Multimodal Pain Program With Telephone Support for Adults With Chronic Temporomandibular Disorder Pain: Pilot Randomized Controlled Trial
Brief Title: An Internet-based Multimodal Pain Program for Chronic Temporomandibular Disorder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Per Alstergren, Professor, Senior Consultant, Pro Dean, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSK2016OFRS01
Record Dates: First submitted 2020-04-20; First posted 2020-04-27 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain; Temporomandibular Disorder
MeSH Terms: conditions — Chronic Pain; Temporomandibular Joint Disorders | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: An unblinded parallel-arm RCT pilot study with equal allocation was conducted. Participants were randomized to the iMPP or to an active control. They were recruited from a general dental care clinic (Fäladstorget) within the National Dental Care Skåne, Sweden. Examination and allocated treatment were free of charge for participants, and no other financial compensation was given. This study is part of a large research project with the primary objective to study changes in the brain after treatment in patients with chronic TMD pain. Therefore, participants went through magnetic resonance imaging (MRI) of the brain pre- and post-treatment. Results from neuroimaging data will be presented elsewhere, however, the feasibility of this additional examination will be addressed here. The study was approved by the Ethics Review Board in Lund, Sweden (No. 2016/6).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The two interventions compared in this study were not possible to blind for the care provider or the patients. Outcome assessment was based on questionnaires why blinding was not considered necessary, although the investigator and outcomes assessor can be regarded as blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based multimodal pain program (Experimental): The iMPP is based on CBT and self-management principles that help patient cope with chronic TMD pain. The iMPP translates a face-to-face therapy to a software platform program.
  Interventions: Behavioral: Internet-based multimodal pain program
- Occlusal splint (Active Comparator): Participants randomized to active control received a hard Michigan-type stabilization splint placed in the upper jaw by one of two calibrated general dentists {Ramfjord, 1994 #276}. The occlusal splint was chosen as the control treatment because it is a conventional and reversible treatment of TMD pain, and it has a known moderate efficacy {Welfare, 2011 #266}.
  Interventions: Device: Occlusal splint

INTERVENTIONS:
Behavioral: Internet-based multimodal pain program — A guided internet-based multimodal pain program for chronic TMD pain
  Other Names: Internet-based cognitive behavioral program
  Arms: Internet-based multimodal pain program
Device: Occlusal splint — Occlusal splint, standard
  Other Names: Michigan splint
  Arms: Occlusal splint

SUMMARY:
Background Chronic temporomandibular disorders (TMD) pain is an undertreated condition in Sweden despite the fact that national guidelines includes effective treatment options. These guidelines recommend multimodal treatment with a behavioral approach. Internet-based intervention is an appealing modality for multimodal TMD treatment, enabling more patients to be reached and treated.

Objective To investigate the treatment effect of an internet-based multimodal pain program (iMPP) on chronic TMD pain. As the study progressed, it also became a measure to evaluate the feasibility of running a larger randomized controlled trial.

DETAILED DESCRIPTION:
BACKGROUND Chronic temporomandibular disorders (TMD) pain is an undertreated condition in Sweden despite the fact that national guidelines includes effective treatment options. These guidelines recommend multimodal treatment with a behavioral approach. Internet-based intervention is an appealing modality for multimodal TMD treatment, enabling more patients to be reached and treated.

Objective To investigate the treatment effect of an internet-based multimodal pain program (iMPP) on chronic TMD pain. As the study progressed, it also became a measure to evaluate the feasibility of running a larger randomized controlled trial.

STUDY DESIGN An unblinded parallel-arm RCT pilot study with equal allocation was conducted. Participants were randomized to the iMPP or to an active control. They were recruited from a general dental care clinic (Fäladstorget) within the National Dental Care Skåne, Sweden. Examination and allocated treatment were free of charge for participants and no other financial compensation was given. This study is part of a large research project with the primary objective to study changes in the brain after treatment in patients with chronic TMD pain. Therefore, participants went through magnetic resonance imaging (MRI) of the brain pre- and post-treatment. The study was approved by the Ethics Review Board in Lund, Sweden (No. 2016/6). This study was not registered in a public trials registry due to its feasibility character.

PARTICIPANTS Participants had to fulfill the following criteria: (1) age between 18 and 75 years; (2) at least one of the TMD pain diagnoses myalgia, myofascial pain with referral, headache attributed to TMD or arthralgia according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) {Schiffman, 2014 #4}; (3) chronic TMD pain (≥3 months), experienced once a week or more often, with an intensity of ≥3 on an 0-10 numeric rating scale (NRS); (4) access to a computer with an internet connection and a mobile phone; (5) sufficient computer literacy and (6) mastery of the Swedish language. Exclusion criteria were: (1) chronic inflammatory systemic disease; (2) all psychiatric disorders except depression and anxiety (due to high comorbidity); (3) occlusal splint therapy in the past 12 months; (4) ongoing extensive dental treatment; and (5) conditions contradicting MRI examination.

Recruitment of participants started in April 2016 and ended in December 2017. Screening was paused during holiday periods (June-August) and during February-April in 2017 due to technical issues with the MRI machine.

PROCEDURE To identify potential participants, all consecutive adult patients visiting for a regular dental check-up were screened. If eligible for the inclusion examination and interested in participation oral and written information about the study was given and a new appointment was booked. The inclusion examination was performed and written informed consent was received. Permuted block randomization with a fixed block size of ten was used. If allocated to iMPP, the participants received working material by mail and the URL to the program was sent by email. Treatment start was assisted by phone. If allocated to treatment with occlusal splint, alginate impressions and index were prepared at the same appointment as the inclusion examination and a new appointment was booked for delivering the splint. Follow-up was performed at three and six months after treatment start by questionnaires sent by mail. Participants also went through an MRI of the brain at baseline (after randomization but before treatment start) and at six months after treatment start at Skåne University Hospital, Malmö, Sweden.

SCREENING The TMD screening tool 2Q/TMD was used to check for initial eligibility {Lövgren, 2016 #293} {Lövgren, 2016 #277}. The screening questions were (Q1) "Do you have pain in your temple, face, jaw or jaw joint once a week or more?" and (Q2) "Do you have pain once a week or more when you open your mouth or chew?". Participants had to answer yes to at least one of the questions and also not fulfill any of the exclusion criteria previously mentioned to be eligible for the inclusion examination.

INCLUSION EXAMINATION All participants underwent a standardized examination according to the DC/TMD to control for eligibility and to collect baseline data. The DC/TMD includes a clinical examination and questionnaires described below {Schiffman, 2014 #4}. Demographic data and pre-treatment expectancies on allocated treatment were also assessed.

CLINICAL EXAMINATION The clinical DC/TMD examination comprises a standardized assessment of pain and headache locations, mouth opening capacity, pain on mandibular movement, pain on palpation, including the presence of referred pain on palpation and temporomandibular joint noises. The clinical examinations were carried out by one of two general dentists calibrated by the DC/TMD Training and Calibration Center at Malmö University, Sweden {Vilanova, 2015 #1}. Re-calibration of the dentists was performed mid-way through the recruitment phase.

The DC/TMD Symptom Questionnaire was used to assess pain symptoms involving the jaw, jaw noise and locking and headache. Data from this questionnaire were combined with the findings in the clinical examination for diagnosis according to DC/TMD {Schiffman, 2014 #4}.

QUESTIONNAIRES Pain The Graded Chronic Pain Scale was used to assess the subdomains characteristic pain intensity (CPI; mean of pain intensity for reported worst, current and average pain) and pain-related disability (DS; mean of how much facial pain changed the patient's ability to participate in daily activities, social activities and work). The questionnaire includes the assessment of pain intensity and pain-related disability that are scored on a 0-10 NRS (modified from{Von Korff, 2011 #279}).

A full-body pain drawing was used to assess pain locations and distribution {Pain, 2020 #278}. The pain distribution was categorized as local (in face area), (iii) regional pain (pain in the neck area in addition to local pain) and (iv) widespread pain (pain at any other site of the body in addition to local or regional pain.

Physical functioning The Jaw Functional Limitation Scale (JLFS-8) was used to assess the overall functional limitation of the masticatory system {Ohrbach, 2008 #280}. The Oral Behaviors Checklist was used to assess the self-reported frequency of oral parafunctional behaviors during awake time {Markiewicz, 2006 #281}.

Emotional functioning The Patient Health Questionnaire was used to assess depression and the Patient Health Questionnaire-15 was used to assess non-specific physical symptoms {Kroenke, 2001 #282}{Kroenke, 2002 #283}. Anxiety was assessed with the Generalized Anxiety Disorders Assessment-7 {Spitzer, 2006 #285}. Stress was assessed with the Perceived Stress Scale-10 and the Pain Catastrophizing Scale was used to assess catastrophizing {Nordin, 2013 #286}{Sullivan, 1995 #287}.

Patient outcome expectancy A Swedish translation of the Stanford Expectations of Treatment Scale (SETS) was used to assess pre-treatment expectancies on allocated treatment {Younger, 2012 #288}.

TREATMENT ARMS INTERVENTION The iMPP is based on CBT and self-management principles that help patient cope with chronic TMD pain. It was developed by orofacial pain specialists at the Department of Orofacial Pain and Jaw Function, Malmö University, Sweden, in collaboration with Psykologpartners AB (a Swedish supplier of internet-based psychological treatment).

The iMPP translates a face-to-face therapy to a software platform program. It can be reached through an URL wherever an internet connection is available and access requires a 2-factor authentication system. A paper-back workbook with homework assignments is included in addition to the internet program. The iMPP consists of seven treatment modules; each described in Table 1 and print screens of the program is shown in Figure 1. Recurrent in each module was a rating of pain frequency, stress levels and life satisfaction to keep track of progression (Fig. 1). Seven weeks was the intended treatment duration: 1 module/week; 40 min/module online plus time for homework assignments. However, access to the program was not time-limited in this pilot study.

The iMPP was designed to be used without HCP involvement, however, in this study, guidance was included in order to increase adherence. A dentist (JL) provided a start-up phone call, follow-up phone calls after each finished module and also sent reminders if necessary. The dentist was also available for additional support through the chat function in the program (asynchronous). At the start-up phone call, participants were guided through the functions in the program and informed about time requirements for the treatment. Follow-up phone calls involved individualized support and feedback; and if participants were unreachable at scheduled follow-up calls, a message through the chat function was sent with the prompt to get in touch. The dentist who guided the treatment had received a 2-day training on internet-based CBT treatment arranged by Psykologpartners AB.

CONTROL CONDITION Participants randomized to active control received a hard Michigan-type stabilization splint placed in the upper jaw by one of two calibrated general dentists {Ramfjord, 1994 #276}. The splints were made of acrylic, covered all the maxillary teeth and had a smooth flat surface. Within 2-6 weeks after treatment start, a check-up appointment was booked. At this check-up appointment, the splint was controlled and, if needed, adjusted. Participants were also encouraged to continue using it.

FOLLOW-UP Follow-up was performed with questionnaires comprising a short version of the DC/TMD axis II instruments.

OUTCOME MEASURES PRELIMINARY EVALUATION OF PARTICIPANT RESPONSES TO INTERVENTION Measures specific to TMD included in the DC/TMD were used as outcome measures, as guided by the Initiative on Methods, Measurement and Pain Assessment in Clinical Trials (IMMPACT). Primary outcomes included characteristic pain intensity, pain-related disability and physical functioning (CPI, DS and JFLS-8). Secondary outcomes were depression and anxiety as measures of emotional functioning. In addition to the IMMPACT core domains, catastrophizing and stress were evaluated as secondary outcomes.

FEASIBILITY Evaluation of the feasibility of the study concerned testing the study protocol and estimation of recruitment and attrition rates in the current research setting. With preliminary results, a post hoc power and sample size calculation were performed. With knowledge of recruitment and attrition rate together with a new estimated sample size, a decision of the feasibility of performing future larger RCT could be taken. The usage metrics of iMPP were not assessed.

ADVERSE EFFECTS Adverse events for iMPP treatment were collected through the follow-up phone calls. Also, all participants randomized to iMPP were given written information at the 3-month follow-up about the opportunity to withdraw from the study and receive rescue treatment if symptoms worsened or they were not satisfied with treatment outcome.

STATISTICAL ANALYSIS Non-parametric statistics were used due to the characteristics of the pain-related variables. Post-hoc power analysis with CPI as the outcome measure was performed. The sample size required for a parametric test on between-group comparison was computed and then 15% additional subjects were added since non-parametric testing will be used in a future RCT {GraphPad Software, 2020 #289}.

Estimation of required sample size was based on a previous neuroimaging study to detect statistically significant results in functional MRI {Gracely, 2002 #290}. According to this, 20 participants in each group should be recruited.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* at least one of the TMD pain diagnoses myalgia, myofascial pain with referral, headache attributed to TMD, or arthralgia according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) {Schiffman, 2014 #4}
* chronic TMD pain (≥3 months), experienced once a week or more often, with an intensity of ≥3 on an 0-10 numeric rating scale (NRS)
* access to a computer with an internet connection and a mobile phone
* sufficient computer literacy and (6) mastery of the Swedish language

Exclusion Criteria:

* chronic inflammatory systemic disease
* all psychiatric disorders except depression and anxiety (due to high comorbidity)
* occlusal splint therapy in the past 12 months
* ongoing extensive dental treatment; and (5) conditions contradicting MRI examination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in The Graded Chronic Pain Scale | 3 months and 6 months follow-ups
  Measures specific to TMD were used as outcome measures, as guided by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations on core domains {Turk, 2003 #300}{Haythornthwaite, 2010 #301}. Primary outcomes included characteristic pain intensity as assessed by the Graded Chronic Pain Scale
Change in Pain-related disability | 3 months and 6 months follow-ups
  Measures specific to TMD were used as outcome measures, as guided by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations on core domains {Turk, 2003 #300}{Haythornthwaite, 2010 #301}. Primary outcomes included pain-related disability assessed bi the Graded Chronic Pain Scale.

SECONDARY OUTCOMES:
Depression | 3 months and 6 months follow-ups
  Degree of depression as a measure of emotional functioning, assessed by the Patient Health Questionnaire-9
Anxiety | 3 months and 6 months follow-ups
  Degree of anxiety as a measure of emotional functioning, assessed by the Generalized Anxiety Disorder-7 questionnaire
Catastrophizing | 3 months and 6 months follow-ups
  Degree of catastrophizing as a measure of emotional functioning, assessed by the Pain Catastrophizing Scale-10
The Patient Stress Scale-10 | 3 months and 6 months follow-ups
  Degree of stress as a measure of emotional functioning, assessed by the Patient Stress Scale-10

CONTACTS AND LOCATIONS:
Overall Officials: Per Alstergren, Professor, Principal Investigator — Malmo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam J, Svensson P, Alstergren P. Internet-Based Multimodal Pain Program With Telephone Support for Adults With Chronic Temporomandibular Disorder Pain: Randomized Controlled Pilot Trial. J Med Internet Res. 2020 Oct 13;22(10):e22326. doi: 10.2196/22326. PMID 33048053